CLINICAL TRIAL: NCT00285597
Title: Ursodeoxycholic Acid Therapy in Chronic Heart Failure: A Placebo-controlled Study Evaluating the Effects of Ursodeoxycholic Acid on Peripheral Blood Flow and Immune Function
Brief Title: Ursodeoxycholic Acid in Chronic Heart Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Heart and Lung Institute (Other)
Collaborators: Dr. Falk Pharma GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02-080
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid

SUMMARY:
This is a double-blind, placebo-controlled, cross-over study evaluating the effects of UDCA on peripheral blood flow and immune function in patients with stable chronic heart failure (CHF). Sixteen patients with CHF will be recruited from the heart failure clinic at the Royal Brompton Hospital. Following baseline evaluation, patients will be randomised to receive either placebo or UDCA at a dose of 1000 mg/day for a period of four weeks. They will then undergo repeat evaluation (peripheral blood flow and immune function). A four week washout period will then take place before the patients cross-over to receive the respective other therapy for a further four weeks (i.e. those first receiving placebo will go onto receive UDCA and vice versa). The study will be completed after a total of twelve weeks, with a final assessment (peripheral blood flow and immune function).

ELIGIBILITY:
Inclusion Criteria:

* age >21 years
* of either sex
* the patient is willing and capable of complying with the requirements of this protocol
* the patient has provided written informed consent
* the patient has clinical evidence of chronic heart failure:

  * reduced ejection fraction (≤40%) or left ventricular impairment on echocardiography (LVEDD ≥60mm)
  * stable clinical condition and medication for at least 1 month prior to the study (New York Heart Association class II-IV).
  * the patient is receiving appropriate conventional medical therapy for heart failure (ACE inhibitor or angiotensin II blocker, diuretics, beta-blocker as indicated and tolerated).

Exclusion Criteria:

* congenital heart disease
* any life-threatening disease, other than heart failure
* active malignancy of any type, or history of a malignancy within previous 5 years. Patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years prior to study enrolment are acceptable.
* previous heart transplant
* severe neuro-muscular disease
* history of unstable angina, myocardial infarction or stroke within 3 months prior to the study
* pregnancy or women of child-bearing age
* treatment with immunosuppressive therapy e.g. steroids for rheumatoid arthritis or obstructive lung disease
* significant renal dysfunction (serum creatinine >250mmol/l), severe liver disease (liver function tests > 3 times normal)
* unable to understand and comply with protocol or to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2006-01

PRIMARY OUTCOMES:
peripheral blood flow as assessed by venous occlusion plethysmography

SECONDARY OUTCOMES:
peak and resting arm and leg post-ischaemic blood flow as assessed by venous occlusion plethysmography
tumor Necrosis Factor-alpha (TNF), sCD14, soluble TNF-Receptor 1, Lipopolysaccharide levels
cellular immune function
endothelin-1, B type natriuretic peptide, E-selectin plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Poole-Wilson, MD, Principal Investigator — National Heart and Lung Institute, Dovehouse Street, London SW3 6LY, UK
Locations (1):
- National Heart and Lung Institute, London, United Kingdom

REFERENCES:
- [Derived] von Haehling S, Schefold JC, Jankowska EA, Springer J, Vazir A, Kalra PR, Sandek A, Fauler G, Stojakovic T, Trauner M, Ponikowski P, Volk HD, Doehner W, Coats AJ, Poole-Wilson PA, Anker SD. Ursodeoxycholic acid in patients with chronic heart failure: a double-blind, randomized, placebo-controlled, crossover trial. J Am Coll Cardiol. 2012 Feb 7;59(6):585-92. doi: 10.1016/j.jacc.2011.10.880. PMID 22300693